CLINICAL TRIAL: NCT00574795
Title: A Phase 3, Open-Label Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants in Japan
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine in Healthy Japanese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3003
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-06

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: 13vPnC — "First dose during 2 to 6 months of age Second dose at least 28 days after the first dose Third dose at least 28 days after the second dose Forth dose during 12 to 15 months of age"

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of the 13-valent pneumococcal conjugate vaccine (13vPnC) in infants of Japanese descent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2 to 6 month-old infant
* Available for entire study period

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal vaccine.
* Previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with a pneumococcal conjugate vaccine.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate any type of injection.
* Known or suspected immune deficiency or suppression.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (17):
- Japan (17):
  - Nagoya, Aichi-ken
  - Toyohashi, Aichi-ken
  - Chiba, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Maebaru-shi, Fukuoka
  - Asahikawa-shi, Hokkaido
  - Sapporo, Hokkaido
  - Yokohama, Kanagawa
  - Yokosuka-shi, Kanagawa
  - Nangoku-shi, Kochi
  - Ise-shi, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi-shi, Mie-ken
  - Kurashiki-shi, Okayama-ken
  - Meguro-ku, Tokyo
  - Setagaya-ku, Tokyo

REFERENCES:
- [Derived] Togashi T, Yamaji M, Thompson A, Giardina PC, Aizawa M, Patterson S, Gruber WC, Scott DA; 3003 Study Group. Immunogenicity and safety of a 13-valent pneumococcal conjugate vaccine in healthy infants in Japan. Pediatr Infect Dis J. 2013 Sep;32(9):984-9. doi: 10.1097/INF.0b013e318293007e. PMID 23538524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Japan from September 2007 to February 2008.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 2, 4, 6 months (infant series) and 12-15 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC
Started | 193
Vaccinated Dose 1 | 193
Vaccinated Dose 2 | 190
Vaccinated Dose 3 | 190
Completed | 188
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 1
Period: After Infant Series
Arm/Group | 13vPnC
Started | 188
Completed | 185
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Period: Toddler Dose
Arm/Group | 13vPnC
Started | 185
Completed | 184
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 13vPnC
Number analyzed (Participants) | 193
Age Continuous [Mean (Standard Deviation); unit: months] | 3.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥ 0.35 μg/mL in the 13vPnC Group After the 3-Dose Infant Series
Description: Percentages of participants achieving World Health Organization (WHO) predefined antibody threshold ≥ 0.35 μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one month after 3-dose infant series (at 7 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After Infant Series: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 2, 4, 6 months (infant series).
Arm/Group | 13vPnC After Infant Series
Number analyzed (Participants) | 176
percentage of participants
  Common Serotypes - Serotype 4 | 100.0 [97.9 to 100.0]
  Common Serotypes - Serotype 6B | 98.3 [95.1 to 99.6]
  Common Serotypes - Serotype 9V | 100.0 [97.9 to 100.0]
  Common Serotypes - Serotype 14 | 100.0 [97.9 to 100.0]
  Common Serotypes - Serotype 18C | 100.0 [97.9 to 100.0]
  Common Serotypes - Serotype 19F | 97.2 [93.5 to 99.1]
  Common Serotypes - Serotype 23F | 97.7 [94.3 to 99.4]
  Additional Serotypes - Serotype 1 | 100.0 [97.9 to 100.0]
  Additional Serotypes - Serotype 3 | 100.0 [97.9 to 100.0]
  Additional Serotypes - Serotype 5 | 100.0 [97.9 to 100.0]
  Additional Serotypes - Serotype 6A | 100.0 [97.9 to 100.0]
  Additional Serotypes - Serotype 7F | 100.0 [97.9 to 100.0]
  Additional Serotypes - Serotype 19A | 100.0 [97.9 to 100.0]

2. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were collected using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 7 days after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 2 months of age (infant series Dose 1).
- 13vPnC Dose 2: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 4 months of age (infant series Dose 2).
- 13vPnC Dose 3: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 6 months of age (infant series Dose 3).
- 13vPnC Toddler Dose: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 12-15 months of age (toddler dose).
Arm/Group | 13vPnC Dose 1 | 13vPnC Dose 2 | 13vPnC Dose 3 | 13vPnC Toddler Dose
Number analyzed (Participants) | 193 | 190 | 190 | 185
percentage of participants
  Tenderness - Any (n=165,156,147,143) | 13.3 | 19.9 | 14.3 | 18.2
  Tenderness - Significant (n=160,152,143,132) | 0.6 | 0.0 | 0.0 | 0.0
  Swelling - Any (n=176,173,165,163) | 47.2 | 53.8 | 53.9 | 57.1
  Swelling - Mild (n=174,171,163,154) | 46.0 | 49.1 | 50.3 | 44.2
  Swelling - Moderate (n=167,164,150,151) | 14.4 | 28.7 | 29.3 | 36.4
  Swelling - Severe (n=160,153,143,132) | 0.0 | 1.3 | 0.7 | 2.3
  Redness - Any (n=186,180,171,166) | 74.2 | 74.4 | 67.8 | 68.1
  Redness - Mild (n=183,179,162,156) | 68.3 | 64.8 | 55.6 | 53.8
  Redness - Moderate (n=170,168,157,155) | 24.7 | 43.5 | 38.9 | 40.6
  Redness - Severe (n=160,153,143,132) | 0.0 | 1.3 | 0.7 | 1.5

3. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever ≥ 37.5 degrees Celsius [C], fever ≥ 38 C but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased appetite, irritability, increased sleep, decreased sleep, hives, use of medication to treat symptoms, and use of medication to prevent symptoms) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after each dose
Population: The safety population included all subjects who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Dose 1: Subjects received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 2 months of age (infant series Dose 1).
- 13vPnC Dose 2: Subjects received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 4 months of age (infant series Dose 2).
- 13vPnC Dose 3: Subjects received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 6 months of age (infant series Dose 3).
- 13vPnC Toddler Dose: Subjects received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 12-15 months of age (toddler dose).
Arm/Group | 13vPnC Dose 1 | 13vPnC Dose 2 | 13vPnC Dose 3 | 13vPnC Toddler Dose
Number analyzed (Participants) | 193 | 190 | 190 | 185
percentage of participants
  Fever ≥37.5°C (n=170,163,154,150) | 32.9 | 33.1 | 40.3 | 50.7
  Fever ≥38°C but ≤39°C (n=163,156,146,137) | 6.7 | 12.2 | 10.3 | 20.4
  Fever >39°C but ≤40°C (n=161,153,143,133) | 1.2 | 2.6 | 2.8 | 5.3
  Fever >40°C (n=160,152,143,132) | 0.0 | 0.7 | 0.0 | 0.0
  Decreased appetite (n=163,158,144,138) | 11.7 | 16.5 | 9.7 | 18.1
  Irritability (n=170,166,149,140) | 30.6 | 36.1 | 23.5 | 26.4
  Increased sleep (n=175,160,153,139) | 40.6 | 29.4 | 22.2 | 24.5
  Decreased sleep (n=169,160,145,138) | 21.3 | 23.1 | 15.9 | 12.3
  Hives (n=160,152,143,132) | 1.3 | 1.3 | 0.7 | 0.0
  Medication to treat symptoms (n=160,153,145,135) | 1.9 | 6.5 | 5.5 | 8.1
  Medication to prevent symptoms (n=160,153,144,134) | 0.6 | 3.3 | 2.1 | 3.0

4. Secondary Outcome: Geometric Mean Antibody Concentration (GMC) in 13vPnC Group Relative After the 3-Dose Infant Series
Description: GMC as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one mone month after 3-dose infant series (at 7 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC After Infant Series
Number analyzed (Participants) | 176
μg/mL
  Common Serotypes - Serotype 4 | 6.76 [6.02 to 7.59]
  Common Serotypes - Serotype 6B | 4.77 [4.07 to 5.59]
  Common Serotypes - Serotype 9V | 3.39 [3.03 to 3.78]
  Common Serotypes - Serotype 14 | 14.69 [13.26 to 16.26]
  Common Serotypes - Serotype 18C | 3.68 [3.27 to 4.14]
  Common Serotypes - Serotype 19F | 5.71 [4.90 to 6.65]
  Common Serotypes - Serotype 23F | 2.57 [2.21 to 3.00]
  Additional Serotypes - Serotype 1 | 5.11 [4.48 to 5.82]
  Additional Serotypes - Serotype 3 | 2.87 [2.55 to 3.24]
  Additional Serotypes - Serotype 5 | 3.85 [3.42 to 4.33]
  Additional Serotypes - Serotype 6A | 3.77 [3.35 to 4.25]
  Additional Serotypes - Serotype 7F | 5.78 [5.19 to 6.45]
  Additional Serotypes - Serotype 19A | 6.97 [6.25 to 7.77]

5. Secondary Outcome: Percentage of Participants Achieving Antibody Level ≥ 0.35 μg/mL in the 13vPnC Group After the Toddler Dose
Description: as for outcome 1
Time Frame: one month after the toddler dose (at 12 - 15 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After Toddler Dose: Participants received one single 0.5mL dose of 13vPnC at 12-15 months of age (toddler dose)
Arm/Group | 13vPnC After Toddler Dose
Number analyzed (Participants) | 178
percentage of participants
  Common Serotypes - Serotype 4 | 100 [97.9 to 100]
  Common Serotypes - Serotype 6B | 100 [97.9 to 100]
  Common Serotypes - Serotype 9V | 100 [97.9 to 100]
  Common Serotypes - Serotype 14 | 100 [97.9 to 100]
  Common Serotypes - Serotype 18C | 100 [97.9 to 100]
  Common Serotypes - Serotype 19F | 98.9 [96 to 99.9]
  Common Serotypes - Serotype 23F | 98.9 [96 to 99.9]
  Additional Serotypes - Serotype 1 | 100 [97.9 to 100]
  Additional Serotypes - Serotype 3 | 99.4 [96.9 to 100]
  Additional Serotypes - Serotype 5 | 100 [97.9 to 100]
  Additional Serotypes - Serotype 6A | 100 [97.9 to 100]
  Additional Serotypes - Serotype 7F | 100 [97.9 to 100]
  Additional Serotypes - Serotype 19A | 100 [97.9 to 100]

6. Secondary Outcome: Geometric Mean Antibody Concentration (GMC) in 13vPnC Group Relative After the Toddler Dose
Description: as for outcome 4
Time Frame: one month after the toddler dose (at 12-15 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC After Toddler Dose
Number analyzed (Participants) | 178
μg/mL
  Common Serotypes - Serotype 4 | 9.70 [8.43 to 11.17]
  Common Serotypes - Serotype 6B | 14.61 [12.52 to 17.05]
  Common Serotypes - Serotype 9V | 4.49 [4.00 to 5.06]
  Common Serotypes - Serotype 14 | 16.33 [14.49 to 18.41]
  Common Serotypes - Serotype 18C | 6.09 [5.34 to 6.95]
  Common Serotypes - Serotype 19F | 12.20 [10.37 to 14.35]
  Common Serotypes - Serotype 23F | 6.55 [5.53 to 7.75]
  Additional Serotypes - Serotype 1 | 9.85 [8.62 to 11.27]
  Additional Serotypes - Serotype 3 | 2.06 [1.83 to 2.32]
  Additional Serotypes - Serotype 5 | 7.31 [6.52 to 8.20]
  Additional Serotypes - Serotype 6A | 11.03 [9.69 to 12.55]
  Additional Serotypes - Serotype 7F | 8.31 [7.39 to 9.35]
  Additional Serotypes - Serotype 19A | 15.97 [14.07 to 18.13]

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series; 13vPnC Post-Infant Series: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at approximately 2, 4, 6 months (infant series).
- 13vPnC Toddler Dose: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 12-15 months (toddler dose).
Arm/Group | 13vPnC Infant Series | 13vPnC Post-Infant Series | 13vPnC Toddler Dose
Serious Adverse Events (participants affected / at risk) | 9/193 | 14/193 | 1/185
Other Adverse Events (participants affected / at risk) | 192/193 | 19/193 | 171/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=193) | 13vPnC Post-Infant Series (N=193) | 13vPnC Toddler Dose (N=185)
Adenovirus infection (Infections and infestations) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Exanthema subitum (Infections and infestations) | 1 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Pertussis (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=193) | 13vPnC Post-Infant Series (N=193) | 13vPnC Toddler Dose (N=185)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pulmonary valve stenosis (Cardiac disorders) | 1 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 2 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0 | 2
Conjunctivitis (Eye disorders) | 16 | 0 | 8
Eye discharge (Eye disorders) | 3 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 32 | 0 | 12
Constipation (Gastrointestinal disorders) | 7 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 163 | 0 | 115
Injection site swelling (General disorders) | 121 | 0 | 94
Pyrexia (General disorders) | 108 | 0 | 80
Irritability (General disorders) | 93 | 0 | 38
Injection site pain (General disorders) | 49 | 0 | 27
Injection site induration (General disorders) | 16 | 0 | 2
Injection site eczema (General disorders) | 0 | 0 | 1
Injection site mass (General disorders) | 3 | 0 | 1
Injection site irritation (General disorders) | 1 | 0 | 0
Injection site warmth (General disorders) | 1 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0
Vaccination site induration (General disorders) | 1 | 0 | 0
Vessel puncture site reaction (General disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
Food allergy (Immune system disorders) | 3 | 8 | 0
Milk allergy (Immune system disorders) | 1 | 0 | 0
Solvent sensitivity (Immune system disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 77 | 0 | 42
Nasopharyngitis (Infections and infestations) | 41 | 0 | 15
Bronchitis (Infections and infestations) | 24 | 1 | 12
Exanthema subitum (Infections and infestations) | 24 | 0 | 7
Gastroenteritis (Infections and infestations) | 19 | 0 | 5
Influenza (Infections and infestations) | 9 | 0 | 1
Pharyngitis (Infections and infestations) | 9 | 0 | 8
Varicella (Infections and infestations) | 9 | 0 | 1
Rhinitis (Infections and infestations) | 7 | 0 | 3
Enteritis infectious (Infections and infestations) | 5 | 0 | 1
Otitis media (Infections and infestations) | 5 | 1 | 10
Otitis media acute (Infections and infestations) | 5 | 0 | 4
Bronchiolitis (Infections and infestations) | 4 | 0 | 1
Croup infectious (Infections and infestations) | 4 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 0 | 4
Molluscum contagiosum (Infections and infestations) | 4 | 0 | 1
Adenovirus infection (Infections and infestations) | 3 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 3 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 2 | 0 | 0
Fungal skin infection (Infections and infestations) | 2 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Skin candida (Infections and infestations) | 2 | 0 | 0
Viral rash (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Enterocolitis viral (Infections and infestations) | 1 | 0 | 0
Enterovirus infection (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 2
Laryngitis (Infections and infestations) | 1 | 0 | 0
Omphalitis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Pertussis (Infections and infestations) | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0
Rotavirus infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1
Herpangina (Infections and infestations) | 0 | 0 | 4
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 47 | 0 | 25
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 101 | 0 | 34
Crying (Nervous system disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 66 | 0 | 17
Head banging (Psychiatric disorders) | 1 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 0 | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 7
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 27 | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 24 | 0 | 10
Rash (Skin and subcutaneous tissue disorders) | 14 | 0 | 1
Eczema infantile (Skin and subcutaneous tissue disorders) | 8 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 6 | 0 | 8
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 22/165 | 0 | 26/143 — Dose 1 Infant Series and Toddler Dose
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 31/156 | 0 | 0 — Dose 2 Infant Series
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 21/147 | 0 | 0 — Dose 3 Infant Series
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 1/160 | 0 | 0/132 — Dose 1 Infant Series and Toddler Dose
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 0/152 | 0 | 0 — Dose 2 Infant Series
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 0/143 | 0 | 0 — Dose 3 Infant Series
Induration (Any) (Skin and subcutaneous tissue disorders) | 83/176 | 0 | 93/163 — Dose 1 Infant Series and Toddler Dose
Induration (Any) (Skin and subcutaneous tissue disorders) | 93/173 | 0 | 0 — Dose 2 Infant Series
Induration (Any) (Skin and subcutaneous tissue disorders) | 89/165 | 0 | 0 — Dose 3 Infant Series
Induration(Mild) (Skin and subcutaneous tissue disorders) | 80/174 | 0 | 68/154 — Dose 1 Infant Series and Toddler Dose
Induration(Mild) (Skin and subcutaneous tissue disorders) | 84/171 | 0 | 0 — Dose 2 Infant Series
Induration(Mild) (Skin and subcutaneous tissue disorders) | 82/163 | 0 | 0 — Dose 3 Infant Series
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 24/167 | 0 | 55/151 — Dose 1 Infant Series and Toddler Dose
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 47/164 | 0 | 0 — Dose 2 Infant Series
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 44/150 | 0 | 0 — Dose 3 Infant Series
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/160 | 0 | 3/132 — Dose 1 Infant Series and Toddler Dose
Induration (Severe) (Skin and subcutaneous tissue disorders) | 2/153 | 0 | 0 — Dose 2 Infant Series
Induration (Severe) (Skin and subcutaneous tissue disorders) | 1/143 | 0 | 0 — Dose 3 Infant Series
Erythema (Any) (Skin and subcutaneous tissue disorders) | 138/186 | 0 | 113/166 — Dose 1 Infant Series and Toddler Dose
Erythema (Any) (Skin and subcutaneous tissue disorders) | 134/180 | 0 | 0 — Dose 2 Infant Series
Erythema (Any) (Skin and subcutaneous tissue disorders) | 116/171 | 0 | 0 — Dose 3 Infant Series
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 125/183 | 0 | 84/156 — Dose 1 Infant Series and Toddler Dose
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 116/179 | 0 | 0 — Dose 2 Infant Series
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 90/162 | 0 | 0 — Dose 3 Infant Series
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 42/170 | 0 | 63/155 — Dose 1 Infant Series and Toddler Dose
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 73/168 | 0 | 0 — Dose 2 Infant Series
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 61/157 | 0 | 0 — Dose 3 Infant Series
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/160 | 0 | 2/132 — Dose 1 Infant Series and Toddler Dose
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 2/153 | 0 | 0 — Dose 2 Infant Series
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 1/143 | 0 | 0 — Dose 3 Infant Series
Any fever (≥37.5°C) (General disorders) | 56/170 | 0 | 76/150 — Dose 1 Infant Series and Toddler Dose
Any fever (≥37.5°C) (General disorders) | 54/163 | 0 | 0 — Dose 2 Infant Series
Any fever (≥37.5°C) (General disorders) | 62/154 | 0 | 0 — Dose 3 Infant Series
Fever ≥38°C but ≤39°C (mild) (General disorders) | 11/163 | 0 | 28/137 — Dose 1 Infant Series and Toddler Dose
Fever ≥38°C but ≤39°C (mild) (General disorders) | 19/156 | 0 | 0 — Dose 2 Infant Series
Fever ≥38°C but ≤39°C (mild) (General disorders) | 15/146 | 0 | 0 — Dose 3 Infant Series
Fever >39°C but ≤40°C (moderate) (General disorders) | 2/161 | 0 | 7/133 — Dose 1 Infant Series and Toddler Dose
Fever >39°C but ≤40°C (moderate) (General disorders) | 4/153 | 0 | 0 — Dose 2 Infant Series
Fever >39°C but ≤40°C (moderate) (General disorders) | 4/143 | 0 | 0 — Dose 3 Infant Series
Fever >40°C (severe) (General disorders) | 0/160 | 0 | 0/132 — Dose 1 Infant Series and Toddler Dose
Fever >40°C (severe) (General disorders) | 1/152 | 0 | 0 — Dose 2 Infant Series
Fever >40°C (severe) (General disorders) | 0/143 | 0 | 0 — Dose 3 Infant Series
Decreased appetite (General disorders) | 19/163 | 0 | 25/138 — Dose 1 Infant Series and Toddler Dose
Decreased appetite (General disorders) | 26/158 | 0 | 0 — Dose 2 Infant Series
Decreased appetite (General disorders) | 14/144 | 0 | 0 — Dose 3 Infant Series
Irritability (General disorders) | 52/170 | 0 | 37/140 — Dose 1 Infant Series and Toddler Dose
Irritability (General disorders) | 60/166 | 0 | 0 — Dose 2 Infant Series
Irritability (General disorders) | 35/149 | 0 | 0 — Dose 3 Infant Series
Increased sleep (General disorders) | 71/175 | 0 | 34/139 — Dose 1 Infant Series and Toddler Dose
Increased sleep (General disorders) | 47/160 | 0 | 0 — Dose 2 Infant Series
Increased sleep (General disorders) | 34/153 | 0 | 0 — Dose 3 Infant Series
Decreased sleep (General disorders) | 36/169 | 0 | 17/138 — Dose 1 Infant Series and Toddler Dose
Decreased sleep (General disorders) | 37/160 | 0 | 0 — Dose 2 Infant Series
Decreased sleep (General disorders) | 23/145 | 0 | 0 — Dose 3 Infant Series
Hives (urticaria) (General disorders) | 2/160 | 0 | 0/132 — Dose 1 Infant Series and Toddler Dose
Hives (urticaria) (General disorders) | 2/152 | 0 | 0 — Dose 2 Infant Series
Hives (urticaria) (General disorders) | 1/143 | 0 | 0 — Dose 3 Infant Series

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.